CLINICAL TRIAL: NCT07055191
Title: Prospective Randomized Multicenter Trial Comparing the Efficacy and Safety of the Transoral Endoscopic Thyroidectomy by Vestibular Approach (TOETVA) Versus Anterior Cervical Thyroidectomy (AC)
Brief Title: TOETVA Technique Compared With Anterior Cervical Thyroidectomy (AC) in Terms of Efficacy and Safety
Acronym: THYRORAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022_0509; PHRC-21-0340 (Other Grant/Funding Number: PHRC-N); 2022-A02301-42 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2025-03-03; First posted 2025-07-08 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Lobectomy; Thyroidectomy
Keywords: Endocrinology; thyroidectomy; mini-invasive; TransOral Endoscopic Thyroidectomy by Vestibular Approach (TOETVA); Anterior Cervical thyroidectomy (AC)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transoral Endoscopic Thyroidectomy by Vestibular Approach (TOETVA) (Experimental)
  Interventions: Procedure: Transoral Endoscopic Thyroidectomy by Vestibular Approach
- Anterior Cervical thyroidectomy (AC) (Active Comparator)
  Interventions: Procedure: Anterior Cervical thyroidectomy

INTERVENTIONS:
Procedure: Transoral Endoscopic Thyroidectomy by Vestibular Approach — Transoral Endoscopic Thyroidectomy by Vestibular Approach
  Arms: Transoral Endoscopic Thyroidectomy by Vestibular Approach (TOETVA)
Procedure: Anterior Cervical thyroidectomy — Anterior Cervical thyroidectomy
  Arms: Anterior Cervical thyroidectomy (AC)

SUMMARY:
Nearly 50,000 thyroidectomies are performed in France each year for benign and malignant pathologies. Each one affects the life of the patient and represents, for some, suffering, symbolized by the stigma of the operation. The consequences of these scars vary according to the patient, their experience and their culture. For example, cervicotomies are particularly badly accepted in Asia since they are supposed to interrupt the fertility meridian. In France, increasing attention is being paid to the global management of a person with some disease. As a disease state may be transitory, the medical team must consider the situation "after the illness" and plan a return to normality. In particular, alternative approaches to cervicotomy have been developed, in which the scar is in a less visible location, at the cost of a more extensive dissection. These techniques include the transaxillary approach, the bi-areolar biaxillary approach and the retroauricular approach. Such procedures, initially developed as an endoscopic approach, have become progressively robotically assisted, to help with the ergonomics of the procedure. Even though robotic assistance initially helped to spread use of these techniques, it has, over time, limited them, first because of higher cost, and second because of the high learning curve (50 to 75 cases). Finally, the transaxillary approach, which is the most commonly performed, has an inherent problem due to the decreased visibility of the noble structures on the contralateral side, leading to frequent subtotal resection.

Since 2014, the Transoral Endoscopic Thyroidectomy by Vestibular Approach (TOETVA) has been developed as an alternative to these robot-assisted procedures. Because this technique offers the surgeon similar access to the anatomical structures on both sides of the trachea and makes it possible to identify the noble structures to be preserved, TOETVA is currently undergoing a more widespread use in France and worldwide and more candidates for are being offered the procedure. TOETVA reduces the need for dissection to reach the thyroid gland. Moreover, this procedure does not require any special equipment, even if robotic assistance has been used in transoral thyroidectomy.

Just like the electric light was not developed from the continuous improvement of candles, entirely new approaches are sometimes necessary in surgery. The Scientific Committee of the French Association of Endocrine Surgery is convinced that TOETVA, will become more widely used in France, even if this technique is a major departure from the standard approach. However, it is technically more demanding and must, therefore, be evaluated and supervised. This will require a safety study and a comparison with the current reference procedure, the anterior cervical thyroidectomy (AC). The investigators assume, based on our initial experience, that the use of endoscopic equipment and its magnification will allow good visualization of the noble elements (recurrent nerve and parathyroid glands) and that the complication rate of TOETVA will not be higher than that of the reference approach.

The investigators propose to evaluate, through a prospective randomized study, an innovative endocrine surgical technique that has started to be used worldwide. Although this study is in line with the objectives of an evaluation of the pertinence of care by the health authorities, it would be the first assessment of this innovative surgical technique in thyroid surgery. To our knowledge, after an extensive bibliographic search, no prospective multicenter randomized trial comparing TOETVA to AC has yet been performed, even if many cohorts of patients have been reported to have benefited from this approach6.

In this trial, any change to the quality of life will be extensively evaluated. The use of validated scores to quantify pain and quality of life will provide objective information and make it possible to determine the impact of the presence or absence of a scar.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a surgical indication for lobectomy or thyroidectomy
* Estimated thyroid volume measured by ultrasonography of less than 60 mL
* Nodules suspected to be malignant measuring less than 4 cm
* Patient aged between 18 and 65 years old
* Patient who has benefited from an endocrinological evaluation, with a favorable opinion for TOETVA or AC Patient who understands and accepts the need for follow-up
* Patient who agrees to be included in the study and who signs the informed consent form
* Patient affiliated to a healthcare insurance plan

Exclusion Criteria:

* Patients refusing an alternative to AC or refusing AC
* History of cervical surgery
* Associated parathyroid surgery
* Identification of malignant lymph nodes
* Presence of a severe and evolutive life threatening pathology
* Patients with unstable psychiatric disorder, under supervision or guardianship
* Patient who does not understand French/ is unable to give consent
* Patient not affiliated to a French or European healthcare insurance
* Patient who has already been included in a trial which has a conflict of interests with the present study
* Pregnant or breast-feeding patient
* Patient incarcerated

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 616 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the non-inferiority of TOETVA compared to AC in terms of early postoperative complications (during the first 24 hours) in patients with a surgical indication for lobectomy or total thyroidectomy without associated lymph node procedure. | during the first 24 hours
  The rate of patients with early postoperative complications defined by the occurrence of at least one of the following events within the first 24 hours:
  * Recurrent paralysis, defined by abnormal vocal cord mobility;
  * Hypoparathyroidism: defined by calcium level<80 mg/L and/or parathyroid hormone level<15 pg/mL;
  * Hematoma: defined by the need for additional surgery to drain the hematoma

SECONDARY OUTCOMES:
To compare, between the two surgical approaches (TOETVA vs. AC) in patients with a surgical indication for lobectomy or total thyroidectomy without associated lymph node procedure, the rate of mid-term postoperative complications | within 30 days of surgery
  The rate of patients with mid-term postoperative complications defined by the occurrence of at least one of the following events within the 30 postoperative days:
  * Symptomatic hypocalcemia secondary to hypoparathyroidism: defined by initiation of calcium supplementation;
  * Hematoma: defined by the a revision surgery for hematoma;
  * Infection: defined by revision surgery for infection or the initiation of an antibiotic therapy, apart from perioperative antibiotic prophylaxis for the TOETVA group.
To compare, between the two surgical approaches (TOETVA vs. AC) in patients with a surgical indication for lobectomy or total thyroidectomy without associated lymph node procedure, the quality of life at 1 month after surgery | at 1 month after surgery
  Quality of life scores assessed at 1 month using the 36-Item Short Form Survey (SF-36), the Voice handicap index (VHI) and the Swallowing Impairment Score (SIS) questionnaires.
  SF36: score from 0 to 100. Higher scores mean a better outcome. VHI: score from 0 to 120. Higher scores mean a worse outcome. SIS: score from 0 to 24. Higher scores mean a worse outcome.
To compare, between the two surgical approaches (TOETVA vs. AC) in patients with a surgical indication for lobectomy or total thyroidectomy without associated lymph node procedure, the quality of life at 6 months after surgery | at 6 months after surgery
  Quality of life scores assessed at 6 months using the 36-Item Short Form Survey (SF-36), the Voice handicap index (VHI) and the Swallowing Impairment Score (SIS) questionnaires.
  SF36: score from 0 to 100. Higher scores mean a better outcome. VHI: score from 0 to 120. Higher scores mean a worse outcome. SIS: score from 0 to 24. Higher scores mean a worse outcome.
To compare, between the two surgical approaches (TOETVA vs. AC) in patients with a surgical indication for lobectomy or total thyroidectomy without associated lymph node procedure, the evolution of pain at 1 month after surgery | at 1 month after surgery
  Change in pain at 1 month from baseline (preoperative assessment), assessed using two validated scores: (1) the visual analogue scale (VAS) in five areas (lower lip, chin, jaw, anterior neck, and cervix/back) and during four actions (swallowing, brushing teeth, speaking, and shaving), which is the only one that has been validated for TOETVA and (2) the DN4 (Neuropathic Pain 4 Questions), which is widely used in the literature.
To compare, between the two surgical approaches (TOETVA vs. AC) in patients with a surgical indication for lobectomy or total thyroidectomy without associated lymph node procedure, the evolution of pain at 6 months after surgery | at 6 months after surgery
  Change in pain at 6 months from baseline (preoperative assessment), assessed using two validated scores: (1) the visual analogue scale (VAS) in five areas (lower lip, chin, jaw, anterior neck, and cervix/back) and during four actions (swallowing, brushing teeth, speaking, and shaving), which is the only one that has been validated for TOETVA and (2) the DN4 (Neuropathic Pain 4 Questions), which is widely used in the literature.

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - AP-HP - Hôpital Avicennes, Bobigny
  - Hôpital Franco-Britannique, Levallois-Perret
  - CHU de Lille, Hôpital Huriez, Lille
  - CHU Dupuytren, Limoges
  - CHU de Nantes - Hôtel Dieu, Nantes
  - AP-HP - Hôpital Cochin, Paris
  - Hôpital Lyon Sud, Pierre-Bénite
  - CHU de Poitiers, Poitiers
  - Polyclinique de la Côte Basque Sud, Saint-Jean-de-Luz
  - CHRU de Nancy Brabois, Vandœuvre-lès-Nancy